CLINICAL TRIAL: NCT01139164
Title: Allogeneic Hematopoietic Stem Cell Transplantation With Reduced-Intensity Pre-Transplant Conditioning for the Treatment of High-Risk Hematological Malignancies
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation With Reduced Intensity Pre-transplant Conditioning for the Treatment of High-risk Hematological Malignancies (V3)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely due to low accrual.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101370; HR#19490 (Other: MUSC IRB)
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2016-02

CONDITIONS: Hematological Malignancies
Keywords: high-risk hematological malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — OOS-A regimen; Regimen B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm, non-randomized study (Experimental)
  Interventions: Drug: Regimen A; Drug: Regimen B; Drug: Regimen C

INTERVENTIONS:
Drug: Regimen A — Chronic Lymphocytic Leukemia/ Chronic Prolymphocytic Leukemia, Multiple Myeloma.
Drug: Regimen B — Other malignancies not addressed in A or C
Drug: Regimen C — B-Cell Lymphomas

SUMMARY:
This is study is for patients that have been diagnosed with high-risk hematological malignancies. The main purpose of this study is to confirm previously published results of stem cell transplantation with reduced intensity pre-transplant conditioning. Patients will be assigned to 1 of 3 regimens depending on the patient's diagnosis. Participants will be followed by the transplant team for the remainder of the patient's life. Patient's will visit MUSC daily, then visits will be reduced to frequent visits for up to 6 months. After 6 months, the visits will be reduced more depending on the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* A proven diagnosis of one of the conditions in Table 1.
* Prior therapy including blood or marrow transplant will not exclude patients for reduced intensity transplant.
* Age < 75 years. Pediatric patients are eligible from the ages of 1 month to 18 years if the transplant physician believes that co-morbid conditions significantly increase the risk for a standard transplant regimen.
* HIV antibody negative.
* ECOG performance status 0-3, (or equivalent Karnofsky and Lansky performance scores for patients <18yrs, see appendix 2)
* Availability of an HLA-identical related donor or suitable alternative donor, (≥7/8 allele match at A, B, C and DRB). Syngeneic transplants will not be allowed in this protocol.
* Due to the complexity of the study, all patients prior to enrollment will be assessed by the PI or co-PI.
* Patient with marrow failure states or immune deficiency syndromes undergoing stem cell transplants must be reviewed by one of the investigators to determine eligibility for study.
* Adequate insurance coverage (or financial resources) to cover the costs associated with the patient's transplant and, in the case of patients eligible for cohort C, to cover the costs associated with I 131 Tositumomab treatment.

Exclusion Criteria:

* Active CNS involvement with malignant disease.
* Pregnancy.
* Fertile men or women unwilling to use contraceptive techniques during the study period.
* Creatinine clearance < 30 ml/min.
* Left ventricular ejection fraction <30% or clinical cardiac failure uncontrolled by medical therapy.
* Pulmonary disease requiring supplemental oxygen therapy.
* Patients with estimated life span less than 1 year due to medical illnesses other than the condition being treated on the study.

Donor Selection:

Inclusion Criteria

* Major HLA identical relative or genotypically matched unrelated donor (7-8/8 alleles) .
* Donors must meet the selection criteria as defined by the Foundation for the Accreditation of Cell Therapy (FACT) and will be screened per the American Association of Blood Banks (AABB) guidelines.

Exclusion Criterion

* Positive anti-donor HLA antibody.
* Identical twin.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-06; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stuart, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Regimen A: Regimen A: Chronic Lymphocytic Leukemia/Chronic Prolymphocytic Leukemia/Multiple Myeloma
- Group 2: Regimen B: Other Malignancies not addressed in regimens A and C
- Group 3: Regimen C: B-Cell Lymphomas
Period: Overall Study
Arm/Group | Group 1: Regimen A | Group 2: Regimen B | Group 3: Regimen C
Started | 4 | 67 | 7
Completed | 4 | 65 | 7
Not Completed | 0 | 2 | 0
Not completed — Withdrawn prior to study start | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who were enrolled to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Regimen A | Group 2: Regimen B | Group 3: Regimen C | Total
Number analyzed (Participants) | 4 | 67 | 7 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 44 | 6 | 54
  >=65 years | 0 | 23 | 1 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 24 | 3 | 27
  Male | 4 | 43 | 4 | 51
Region of Enrollment [Number; unit: participants]
  United States | 4 | 67 | 7 | 78

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Treatment-related Mortality Rate of Allogeneic Stem Cell Transplants Using Reduced-intensity Conditioning Regimens Within 1st 100-days.
Description: Number of subject deaths prior to day 100.
Time Frame: 8 years
Population: For regimen B, only the subjects who participated in study intervention were analyzed for outcome measures.
Measure: Number; unit: participants
Arm/Group | Group 1: Regimen A | Group 2: Regimen B | Group 3: Regimen C
Number analyzed (Participants) | 4 | 65 | 7
participants | 0 | 18 | 0

2. Secondary Outcome: To Determine the Engraftment Rate of Allogeneic Stem Cell Transplants
Description: To determine the engraftment rate of allogeneic stem cell transplants using reduced-intensity conditioning regimens. It will be measured as the proportion of subjects meeting criteria for engraftment before day +30 and full donor chimerism demonstrated before or at day +100. Engraftment is defined by maintenance of ANC > 500/mm3 for at least 3 consecutive days and platelet count > 20,000/mm3 for 3 consecutive days in absence of platelet transfusion. These criteria must have been met before Day +30. Chimerism is the pressence of donor cells and will be analyzed by FISH for sex-mismatched donor-recipient pairs and VNTR analysis for sex-mathced pairs. Chimerism by Day +100 will be documented for this outcome
Time Frame: Day +100
Population: The outcome measure data below only accounts for the number of subjects who met the engraftment criteria prior at day +30; the chimerism data was not collected. For regimen B, only the subjects who participated in study intervention were analyzed for outcome measures.
Measure: Number; unit: participants
Arm/Group | Group 1: Regimen A | Group 2: Regimen B | Group 3: Regimen C
Number analyzed (Participants) | 4 | 65 | 7
participants | 3 | 46 | 6

3. Secondary Outcome: Morbidity of Allogeneic Stem Cell Transplants
Description: To determine the morbidity, including the pattern and severity of complications, of allogeneic stem cell transplants using reduced-intensity conditioning regimens. The average number of days spent in the hospital until day +100 will be reported as a surrogate for morbidity and complications.
Time Frame: 100 days
Population: This study terminated early; funding ran out before the analysis could be completed.
Arm/Group | Group 1: Regimen A | Group 2: Regimen B | Group 3: Regimen C
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Start of treatment until end of study
Description: repotable adverse events included:
  any deaths occuring on study, any grade IV non-hematological toxicity until 1 year post transplant or 6 months after the last donor lymphocyte infusion (whichever is latest), severe (grade III or IV) acute graft versus host disease (GVHD) any unexpected adverse events
Arm/Group | Group 1: Regimen A | Group 2: Regimen B | Group 3: Regimen C
Serious Adverse Events (participants affected / at risk) | 0/4 | 32/67 | 0/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/67 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Regimen A (N=4) | Group 2: Regimen B (N=67) | Group 3: Regimen C (N=7)
altered mental status (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
GVHD (Infections and infestations) | 0 (0) | 15 (15) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
anoxic brain damage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
TA-TMA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes